CLINICAL TRIAL: NCT00024284
Title: A Phase I Study Of Carboplatin And Irinotecan In Patients 1-21 Years Of Age With Refractory Solid Tumors
Brief Title: Carboplatin and Irinotecan in Treating Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068908; BMS-CA124-001; CNMC-2782; MSKCC-01071; SJCRH-CARCPT; NCI-G01-2016
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Carboplatin; Irinotecan

INTERVENTIONS:
Drug: carboplatin
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of combining carboplatin and irinotecan in treating children who have refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of carboplatin and irinotecan in children with refractory solid tumors.
* Determine the safety profile and dose-limiting toxic effects of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the preliminary anti-tumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of carboplatin and irinotecan.

Patients receive carboplatin IV over 50 minutes on day 1 and irinotecan IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of carboplatin and irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for at least 30 days.

PROJECTED ACCRUAL: A total of 25-30 patients will be accrued for this study within 6-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor, including primary brain tumor

  * Progressive disease on standard therapy or for which no standard therapy exists
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* 1 to 21

Performance status:

* Lansky 50-100% (age 10 and under)
* Karnofsky 50-100% (over age 10)

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT no greater than 2.5 times upper limit of normal

Renal:

* Glomerular filtration rate at least 30 mL/min

Other:

* No active infection
* No serious uncontrolled medical disorder
* No psychiatric disorder or other disorder that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 6 months since prior allogeneic bone marrow transplantation without evidence of acute or chronic graft versus host disease
* At least 3 months since prior autologous bone marrow or peripheral blood stem cell transplantation
* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunotherapy

Chemotherapy:

* No more than 3 prior chemotherapy regimens
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent hormone replacement therapy or oral contraceptives allowed
* No other concurrent hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy (including for brain metastases) and recovered
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational anticancer drugs
* No other concurrent antitumor therapy
* No concurrent anticonvulsants (e.g., phenytoin, phenobarbital, or carbamazepine) except gabapentin (Neurontin)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2001-06; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Gollerkeri, MD, Study Chair — Bristol-Myers Squibb
Locations (7):
- United States (6):
  - Arizona Cancer Center, Tucson, Arizona
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University Medical Center, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Hospital for Sick Children, Toronto, Ontario, Canada